CLINICAL TRIAL: NCT00758615
Title: Pilot and Feasibility Evaluation of a Walking School Bus Program Intervention for Elementary School Students
Brief Title: Pilot Evaluation of a Walking School Bus Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jason Mendoza, Associate Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21CA133418-01 (NIH); 163773
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Physical Activity; Pedestrian Safety; Injury Prevention
Keywords: Obesity; Physical activity; Injury Prevention; Pedestrian safety; Self efficacy; School; Walking School Bus; Safe Routes to School
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Walking School Bus Intervention
  Interventions: Behavioral: Walking School Bus
- C (No Intervention): Usual school procedures for student transportation to school

INTERVENTIONS:
Behavioral: Walking School Bus — Students are chaperoned to and from school by adults (study staff or parent volunteers) along set routes.
  Other Names: Safe Routes to School
  Arms: I

SUMMARY:
Walking to school is one of the objectives for children and adolescents in Healthy People 2010 and in previous studies was associated with higher levels of overall physical activity, which has been shown to decrease obesity. Therefore, more children walking to school should result in increased physical activity and presumably reduce obesity. However, increasing child pedestrian activity could increase the risk of child pedestrian injuries. Walking with an adult who provides instruction in pedestrian skills and monitors the child's actual behavior may be the most important component of a successful intervention. Walking with an adult reduced child pedestrian injury risk by almost 70%. A walking school bus (WSB) addresses safety concerns by providing a period of physical activity supervised by several responsible adults and teaching opportunities around pedestrian safety skills on the way to and from school. Children may join the WSB at various points along the set route. Despite the growing popularity of WSB programs in the United States, randomized, controlled-studies are lacking that examine the impact on children's safety, physical activity, and health. We seek to help fill this gap in the literature by piloting a WSB program in elementary schools in the Houston Independent School District to test feasibility. We hypothesize that a WSB program will: (1) increase the number of students walking to school and decrease the number of students driven to school by car, (2) increase students' pedestrian safety behaviors (3) increase students' physical activity, and (4) decrease students' excess weight gain.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade student at a study school in the Houston Independent School District
* Must be physically able to walk to and from school

Exclusion Criteria:

* Any condition that would prevent the student from walking to or from school

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Method of student transportation to school | Immediately pre- and post-intervention

SECONDARY OUTCOMES:
Physical activity | Immediately pre- and post-intervention
  Physical activity objectively measured by accelerometers.
Pedestrian crosswalk behavior | Immediately pre- and post-intervention
Parents' psychosocial constructs related to allowing their child to walk to school | Immediately pre- and post-intervention
Child's self-efficacy for walking to school | Immediately pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Mendoza, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Mendoza JA, Watson K, Baranowski T, Nicklas TA, Uscanga DK, Hanfling MJ. The walking school bus and children's physical activity: a pilot cluster randomized controlled trial. Pediatrics. 2011 Sep;128(3):e537-44. doi: 10.1542/peds.2010-3486. Epub 2011 Aug 22. PMID 21859920